CLINICAL TRIAL: NCT01662752
Title: A Study to Assess Near Infrared Laparoscopy With Indocyanine Green (ICG) for Intraoperative Lymphatic Imaging and Sentinel Lymph Node Identification During Standard Surgical Resection for Colonic Cancer
Brief Title: Lymphatic Mapping for Sentinel Node Identification and Analysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C/32/2012
Record Dates: First submitted 2012-08-07; First posted 2012-08-10 (Estimated); Results first posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Colorectal Cancer
Keywords: Early colonic cancer; Sentinel lymph node mapping; Sentinel lymph node biopsy; Near infrared imaging; Indocyanine green; Laparoscopic
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Indocyanine green (Other): Indocyanine green is used for intraoperative identification of sentinel lymph nodes in patients with early colonic cancer using near infrared laparoscopic imaging
  Interventions: Drug: Indocyanine green

INTERVENTIONS:
Drug: Indocyanine green — Please see arm description

SUMMARY:
The main objective of this study is to determine whether the first (sentinel) lymph nodes in the drainage pathway of colonic tumour can be detected at the time of surgery using a new technique. The detection method is to inject a fluorescent dye (indocyanine green) adjacent to the tumour. The dye will then be seen as it fluoresces in the light form the near infrared spectrum that can be used at the time of the laparoscopic (keyhole) surgery. An endoscope is placed in the colon (colonoscopy) during surgery and the tracer fluorescent agent is injected around the tumour. The mesentery in which the lymph nodes draining the tumour are located will then be examined by laparoscopy as it is expected that fluorescence will be identified within approximately 5 minutes of the injection. The first lymph node or nodes that take up the fluorescent dye will then be marked by placing a clip or a stitch by them. After the surgery has been completed and colon removed all lymph nodes can be examined microscopically by the pathologist, paying a particular attention to whether any tumour cells are present in the sentinel lymph nodes and whether the presence or the absence of tumour cells in that node accurately reflects the tumour status of the rest of the specimen.

If this pilot demonstrates that sentinel lymph nodes can be reliably detected, we have developed a technique which allows us to remove a small area (less than 5 cm) of the colon. Using this procedure should decrease complications following traditional surgery. We however also need a method that allows accurate assessment of the lymph nodes draining the tumour. This pilot trial will examine our ability to detect such 'sentinel' lymph nodes so that we can use their status (positive for cancer cells or negative) to determine whether a smaller operation such as full thickness localised excision is adequate treatment for the patient and that they can avoid a larger operation.

DETAILED DESCRIPTION:
Colorectal cancer is the third commonest cancer and second highest cause of cancer death in the United Kingdom (UK). Introduction of the National Bowel Cancer Screening Program and increasing awareness of symptoms of colorectal cancer will lead to an increase in numbers of cancers detected at an early stage of the disease. Standard surgical management, however, remains unchanged and that is segmental colectomy with en bloc mesenteric resection of the regional lymph nodes as the metastatic status of these nodes remains the most important factor for determining adjuvant treatment.

This of course was appropriate when the majority of the patients diagnosed with colorectal cancer presented with symptomatic, locally advanced disease. Our practice, however, needs to be reconsidered in the view of the recently published data from screening centres. Pilot results demonstrate a significant shift towards an earlier stage of the disease in the screened population and suggests that, in future, up to 50% of screen detected-cancers will be T1 or T2 (i.e. early stage disease) 1. Less than 15% of patients with T1 and T2 disease have nodal involvement 2 but current radiological techniques are not sensitive enough to identify these patients pre-operatively. Instead, major surgery is performed in all patients with T1 and T2 stage colonic cancer, and in up to 85%, en bloc mesenteric resection provides no therapeutic benefit, as they have node negative disease. Major resection also exposes patients to a significant risk of morbidity and mortality, along with late side effects.

The concept of sentinel lymph node mapping (SLNM) in colorectal cancer is not new and although it has not had the same impact as in the clinical care of breast cancer, melanoma, and more recently gastric cancer 3-6, some expert centres have suggested that it may be clinically relevant 7, 8. The technique is based on the principle that the first possible sites of metastasis along the lymphatic drainage route from the primary lesion are known as sentinel lymph nodes (SLNs) and these can be detected using injection of dyes, radioisotopes or a combination of both. Therefore, evaluation of the SLNs can result in an accurate assessment of the nodal status in the entire lymphatic basin allowing a tailored surgical treatment. Although this technique has transformed surgical care for melanoma and breast cancer patients, its application in patients with colorectal cancer has been questioned due to discrepancies in the reported results caused by the heterogeneous study designs employed, variations in surgical experience and differing patient inclusion criteria 9-11.

Detailed analysis of studies performed to date shows that tumour and patient characterisation as well as surgeons experience are key factors when assessing the utility of the technique 2, 12 and at least three nodes need to be found in order to maximise this 13. The main research focus so far has been on optimising the technique itself. Initial research was performed using blue dye, radioactive colloid or both in combination but this failed to achieve the 95-97% identification rates found in breast cancer and was also accompanied by unacceptable false negative rates 14-17. Although many authors noted that their false negatives occurred predominantly in patients with advanced disease (T3 and T4 cancers) 18-20, utilisation of those identification agents has proven frustrating to date. Radioactive colloids require involvement of a nuclear medicine physician, can be difficult to localise with a handheld camera and cause signal interference if the SLN(s) is too close to the injection site. Blue dyes however are difficult to localise in patients with a high body mass index (BMI), who unfortunately comprise the majority of our patient population, thus producing only limited (if any) visualisation of afferent lymphatic vessels and SLN(s).

In order to re-examine extensive research that has been reported on SLNM, a secondary intention analysis of the two largest multicentre SLN databases was undertaken. This reported that in 225 patients with T1 or T2 disease, accurate detection of SLNs was possible in 95%, confirming that this staging technique should be most accurate in patients with early colonic cancer 2. This improved with operator experience and when tumour size was smaller than 35 mm in diameter. In 196 patients treated by experienced surgeons, 144 (73.4%), would have correctly undergone localised full thickness resection if surgery had been based only on their SLNs status and 49 (25.0%), would have required conventional resection either because the SLNs were not identified, or due to detection of metastases. Only 3 patients (1.5%) would have been inappropriately predicted to be node negative.

To overcome the aforementioned issues, a number of researchers have utilized optical imaging using the near-infrared (NIR) fluorescence lymphatic tracer indocyanine green (ICG) which enables real-time intraoperative visualisation of lymphatic channels and SLNs. The technique performs as well as the combination of a radioactive tracer and blue dye in patients with breast cancer 21, and has also been validated in patients with early gastric cancer 4-6.

ICG was initially recommended as a tattooing agent for colonic and pancreatic lesions to aid perioperative localization 22-24, as there were no reports of complications such as focal peritonitis, abscess formation, postoperative adhesions and ileus which had been seen with the use of India ink 25-27. However, its use as a tattooing agent is limited to patients undergoing surgery within 8 days after endoscopic injection, as the dye dissipates through lymphatic channels due to its small molecular size 22. More recently, its fluorescence properties have been utilised for intraoperative localisation of colorectal neoplasms and associated SLNs 28-32 in patients undergoing surgery using either charge-coupled device (CCD) or a NIR camera. Nagata et al. demonstrated that observation of ICG dye using a NIR camera was far superior to that by conventional laparoscopy with identification of SLNs being five times better 29. These results suggest that a SLNM technique using NIR with a fluorescent tracer may be useful in patients with a high BMI who have large amounts of mesenteric adipose tissue. All authors reporting the NIR technique have noted its success in colorectal practice, without adverse effects with a comparable role to its use in early breast or gastric cancer.

The ability to utilise this technique and confidently identify the SLNs has the potential to transform the surgical care of patients with colonic neoplasia. The focus, however, must be on patients with early disease, thus allowing those who have node negative disease to be considered for localised full thickness resection of their primary cancer as definitive surgical therapy. Unfortunately, studies published to date have included patients with T3 disease in their series 29, 31.

This pilot trial aims to apply a well-described technique using a NIR camera and ICG as the tracer in order to clarify whether SLNs can be confidently identified in patients undergoing conventional resection (segmental colectomy and en bloc mesenteric resection) for T1 and T2 colonic cancers. This protocol is based on extensive literature search of studies describing the technique in patients with early gastric and colorectal cancers 5, 6, 29-31, 33-36. Provided that the pilot trial is successful, and in order to obtain adequate power, a further large multicentre trial will be required to determine whether the nodes visualised by NIR mapping are representative of the patient's lymphatic basin metastatic status. Proven concordance between the pathology of the SLNs and that of the standard nodal resection would then justify a more limited surgical intervention, taking just the SLN(s), and allowing a more precisely tailored operative intervention.

All patients in the pilot trial will undergo standard surgical treatment in addition to the NIR SLNM technique.

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing and able to give informed consent for participation in the study
2. Patients willing and able to comply with the study procedures
3. Male or Female, aged 18 years or above
4. Patients diagnosed with T1 or T2 colonic neoplasia on preoperative staging and require laparoscopic surgical excision
5. If female, a negative pregnancy test for women of childbearing potential prior to surgery
6. Patients who have clinically acceptable laboratory results pre-operatively with serum creatinine of <110 mg/dL

Exclusion Criteria:

1. Patients diagnosed with T3 or T4 disease on preoperative imaging
2. A patient who is pregnant, lactating or planning pregnancy during the course of the study
3. Allergy to any of the compounds being used for lymphatic mapping including Indocyanine green or sodium iodide
4. Patients with hyperthyroidism or those with thyroid adenomas
5. Patients with renal insufficiency (serum creatinine of >110 mg/dL)
6. Patients in whom the use of ICG is contraindicated including development of adverse events when previously or presently administered
7. Previous allergic reaction to shellfish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin Kennedy, FRCS, MS, Principal Investigator — Imperial College London
Locations (1):
- North West London Hospital, London, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Currie AC, Brigic A, Thomas-Gibson S, Suzuki N, Moorghen M, Jenkins JT, Faiz OD, Kennedy RH. A pilot study to assess near infrared laparoscopy with indocyanine green (ICG) for intraoperative sentinel lymph node mapping in early colon cancer. Eur J Surg Oncol. 2017 Nov;43(11):2044-2051. doi: 10.1016/j.ejso.2017.05.026. Epub 2017 Aug 23. PMID 28919031

RESULTS

PARTICIPANT FLOW:
Groups:
- Indocyanine Green: Single inject a fluorescent dye (indocyanine green) adjacent to the tumour. The dye will then be seen as it fluoresces in the light form the near infrared spectrum that can be used at the time of the laparoscopic (keyhole) surgery. An endoscope is placed in the colon (colonoscopy) during surgery and the tracer fluorescent agent is injected around the tumour. The mesentery in which the lymph nodes draining the tumour are located will then be examined by laparoscopy as it is expected that fluorescence will be identified within approximately 5 minutes of the injection.
Period: Overall Study
Arm/Group | Indocyanine Green
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Indocyanine Green
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16
Region of Enrollment [Number; unit: participants]
  United Kingdom | 30

OUTCOME MEASURES:

1. Primary Outcome: Subjects in Which the SLN(s) Are Identified
Description: To establish whether it is possible to identify the first order draining mesocolic lymph nodes (sentinel lymph node(s) (SLNs) in patients with suspected T1 and T2 colonic cancer, using Indocyanine Green (ICG), a fluorescent mapping agent, and a laparoscopic near infrared imaging (NIR) system
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Indocyanine Green
Number analyzed (Participants) | 30
Participants | 27

2. Secondary Outcome: Sensitivity and Specificity of Tumour-bearing Status of SLN(s) as a Measure of Lymph Node Status When Assessed by Standard Techniques
Description: To assess the extent to which that the tumour-bearing status of SLN(s) identified corresponds with lymph node status as assessed by standard methods (pathological examination of excised nodes using H&E and immunohistochemistry)
Time Frame: 28 days
Population: There were 10 patients with positive nodes hence this is the denominator for the sensitivity analysis. There were 20 patients with negative lymph nodes overall hence this is the denominator for the specificity analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Indocyanine Green
Number analyzed (Participants) | 30
Participants
  Sensitivity: number analyzed (Participants) | 10
  Sensitivity | 3
  Specificity: number analyzed (Participants) | 20
  Specificity | 20

3. Other Pre Specified Outcome: Frequency and Tumour-bearing Status of Aberrant SLN(s
Description: To estimate the proportion of patients with aberrant nodal drainage. i.e. the proportion with SLN(s) lying outside the standard resection field
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Indocyanine Green
Number analyzed (Participants) | 30
Participants | 0

ADVERSE EVENTS:
Time Frame: 2 year
Arm/Group | Indocyanine Green
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 30/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indocyanine Green (N=30)
Wound pain (Injury, poisoning and procedural complications) | 29
Nausea (Gastrointestinal disorders) | 12
Atrial fibrillation (Cardiac disorders) | 1
Dizziness (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Paroxysmal atrial fibrillation (Cardiac disorders) | 1
Bloating (Gastrointestinal disorders) | 2
Constipations (Gastrointestinal disorders) | 1
Distended abdomen (Gastrointestinal disorders) | 1
Epigastric pain (Gastrointestinal disorders) | 1
Hiccough (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 3
Febrile reaction (General disorders) | 1
Rigors (General disorders) | 1
Urinary tract infection (Infections and infestations) | 2
Postoperative ileus (Injury, poisoning and procedural complications) | 1
Low haemoglobin (Investigations) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Tremor (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Low blood pressure (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No